CLINICAL TRIAL: NCT02255500
Title: Evaluation of the Pharmacokinetics and Safety of Local Administration of EXPAREL in Subjects Undergoing Femoral Nerve Block With Bupivacaine HCl for Unilateral Total Knee Arthroplasty
Brief Title: EXPAREL Infiltration in Subjects Undergoing Femoral Nerve Block With Bupivacaine HCl for Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 402-C-406
Record Dates: First submitted 2014-09-23; First posted 2014-10-02 (Estimated); Results first posted 2020-11-24 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-02

CONDITIONS: Pain
Keywords: Total knee arthroplasty
MeSH Terms: conditions — Pain | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bupivacaine FNB + EXPAREL Infiltration (Experimental): Femoral nerve block with bupivacaine HCl 0.5% with epinephrine 1:200,000 within 2 hours of the surgical procedure. Infiltration of EXPAREL 266 mg just prior to wound closure.
  Interventions: Drug: Bupivacaine FNB; Drug: EXPAREL Infiltration

INTERVENTIONS:
Drug: Bupivacaine FNB — A single administration of bupivacaine HCl 0.5% with epinephrine 1:200,000 in 20 mL volume will be administered within 2 hours prior to the surgical procedure as an ultrasound-guided FNB.
  Other Names: Bupivacaine
Drug: EXPAREL Infiltration — A single dose of EXPAREL 266 mg expanded to 60 mL with preservative-free sterile normal saline will be infiltrated into the surgical site just prior to wound closure.
  Other Names: Liposomal bupivacaine

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics of EXPAREL in subjects who undergo femoral nerve block with bupivacaine HCl for unilateral total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
On Day 1, eligible subjects will receive a single 20 mL dose of bupivacaine hydrochloride (HCl) 0.5% with epinephrine 1:200,000 within 2 hours prior to the surgical procedure as an ultrasound-guided femoral nerve block (FNB). EXPAREL 266 mg expanded to 60 mL with preservative-free sterile normal saline will be infiltrated into the surgical site prior to wound closure. There will be no local coadministration of the two drugs.

Blood samples for bupivacaine pharmacokinetic (PK) analysis will be obtained from subjects at baseline (prior to bupivacaine HCl administration for nerve block), 15 minutes, 30 minutes, and 1, 2, 4, 8, 12, 24, 48, 72, and 96 hours after the beginning of EXPAREL administration, and on Day 14.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥18 years of age.
2. American Society of Anesthesiologists (ASA) physical status 1, 2, or 3.
3. Scheduled to undergo femoral nerve block in conjunction with unilateral TKA.
4. Female subjects must be surgically sterile, at least 2 years postmenopausal, or using a medically acceptable method of birth control. Females of childbearing potential must have a documented negative blood or urine pregnancy test result within 24 hours before surgery.
5. Able to provide informed consent, adhere to the study schedule, and complete all study assessments.

Exclusion Criteria:

1. History of hypersensitivity or idiosyncratic reactions to amide-type local anesthetics or opioids.
2. Contraindication to bupivacaine.
3. Received bupivacaine or any other local anesthetic within 7 days of EXPAREL administration.
4. Currently pregnant, nursing, or planning to become pregnant during the study or within 1 month after EXPAREL administration.
5. Planned concurrent surgical procedure (e.g., bilateral TKA).
6. Body weight <50 kg (110 pounds) or a body mass index ≥45 kg/m2.
7. Received any investigational drug within 30 days prior to EXPAREL administration, and/or has planned administration of another investigational product or procedure during the subject's participation in this study.
8. Previous participation in an EXPAREL study.
9. Malignancy in the last 2 years, with the exception of non-metastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
10. Current or historical evidence of any clinically significant disease or condition, especially cardiovascular or neurological conditions that, in the opinion of the Investigator, may increase the risk of surgery or complicate the subject's postsurgical course.
11. Clinically significant medical or psychiatric disease that, in the opinion of the Investigator, would constitute a contraindication to participation in the study, or cause inability to comply with the study requirements.

    In addition, the subject will be ineligible to receive EXPAREL if he or she meets the following criteria during surgery:
12. Any clinically significant event or condition uncovered during the surgery (e.g., excessive bleeding, acute sepsis) that might render the subject medically unstable or complicate the subject's postsurgical course.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Leiman, MD, Principal Investigator — Research Concepts, GP, LLC
Locations (1):
- Research Concepts, GP, LLC, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupivacaine FNB + EXPAREL Infiltration: Femoral nerve block with bupivacaine hydrochloride (HCl) 0.5% with epinephrine 1:200,000 within 2 hours of the surgical procedure. Infiltration of EXPAREL 266 mg just prior to wound closure.
  Bupivacaine FNB: A single administration of bupivacaine HCl 0.5% with epinephrine 1:200,000 in 20 mL volume will be administered within 2 hours prior to the surgical procedure as an ultrasound-guided FNB.
  EXPAREL Infiltration: A single dose of EXPAREL 266 mg expanded to 60 mL with preservative-free sterile normal saline will be infiltrated into the surgical site just prior to wound closure.
- Bupivacaine FNB + EXPAREL Infiltration Admixed With Bupivacaine: Femoral nerve block (FNB) with bupivacaine HCl 0.5% with epinephrine 1:200,000 within 2 hours of the surgical procedure. Infiltration of EXPAREL 266 mg admixed with bupivacaine HCl 0.5% with epinephrine 1:200,000 just prior to wound closure.
  Note: Seven subjects received EXPAREL mixed with bupivacaine with epinephrine. The data for these subjects are summarized as a separate arm from "Bupivacaine FNB + EXPAREL Infiltration."
Period: Overall Study
Arm/Group | Bupivacaine FNB + EXPAREL Infiltration | Bupivacaine FNB + EXPAREL Infiltration Admixed With Bupivacaine
Started | 16 | 7
Completed | 15 | 7
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Bupivacaine FNB + EXPAREL Infiltration: FNB with bupivacaine HCl 0.5% with epinephrine 1:200,000 within 2 hours of the surgical procedure. Infiltration of EXPAREL 266 mg just prior to wound closure.
  Bupivacaine FNB: A single administration of bupivacaine HCl 0.5% with epinephrine 1:200,000 in 20 mL volume will be administered within 2 hours prior to the surgical procedure as an ultrasound-guided FNB.
  EXPAREL Infiltration: A single dose of EXPAREL 266 mg expanded to 60 mL with preservative-free sterile normal saline will be infiltrated into the surgical site just prior to wound closure.
- Total: Total of all reporting groups
Arm/Group | Bupivacaine FNB + EXPAREL Infiltration | Bupivacaine FNB + EXPAREL Infiltration Admixed With Bupivacaine | Total
Number analyzed (Participants) | 16 | 7 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (8.61) | 59.7 (7.04) | 64.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 13 | 7 | 20
  Unknown or Not Reported | 0 | .0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 15 | 6 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 7 | 23

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum observed plasma concentration of a drug in the body after the drug has been administered.
  Blood samples for bupivacaine pharmacokinetic (PK) analysis were to be obtained from subjects at baseline (prior to bupivacaine HCl administration for nerve block), 15 minutes, 30 minutes, and 1, 2, 4, 8, 12, 24, 48, 72, and 96 hours, and 14 days after the beginning of EXPAREL administration
Time Frame: Baseline, 0.25, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, and 96 hours, and 14 days post-dose
Population: The PK analysis set includes all subjects who received bupivacaine HCl with epinephrine and EXPAREL, provided sufficient samples to allow for calculation of the PK parameters required for analysis, and did not have significant protocol deviations that might have invalidated or biased the results.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bupivacaine FNB + EXPAREL Infiltration | Bupivacaine FNB + EXPAREL Infiltration Admixed With Bupivacaine
Number analyzed (Participants) | 14 | 7
ng/mL | 499 (148) | 775 (299)

2. Primary Outcome: Time to Peak Plasma Concentration (Tmax)
Description: The time to reach the maximum observed plasma concentration (Cmax)
  Blood samples for bupivacaine PK analysis were to be obtained from subjects at baseline (prior to bupivacaine HCl administration for nerve block), 15 minutes, 30 minutes, and 1, 2, 4, 8, 12, 24, 48, 72, and 96 hours, and 14 days after the beginning of EXPAREL administration
Time Frame: Baseline, 0.25, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, and 96 hours, and 14 days post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Bupivacaine FNB + EXPAREL Infiltration | Bupivacaine FNB + EXPAREL Infiltration Admixed With Bupivacaine
Number analyzed (Participants) | 14 | 7
hours | 0.675 [0.183 to 78.0] | 47.450 [0.183 to 72.9]

3. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Time of the Last Quantifiable Concentration After Drug Administration (AUC0-last)
Description: Total drug exposure up to the last measurable concentration
  Blood samples for bupivacaine PK analysis were to be obtained from subjects at baseline (prior to bupivacaine HCl administration for nerve block), 15 minutes, 30 minutes, and 1, 2, 4, 8, 12, 24, 48, 72, and 96 hours, and 14 days after the beginning of EXPAREL administration
Time Frame: Baseline, 0.25, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, and 96 hours, and 14 days post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | Bupivacaine FNB + EXPAREL Infiltration | Bupivacaine FNB + EXPAREL Infiltration Admixed With Bupivacaine
Number analyzed (Participants) | 14 | 7
hours*ng/mL | 28234 (10710) | 46600 (16489)

4. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 Extrapolated to Infinity After Drug Administration (AUC0-∞)
Description: Total drug exposure, extrapolated to infinity
  Blood samples for bupivacaine PK analysis were to be obtained from subjects at baseline (prior to bupivacaine HCl administration for nerve block), 15 minutes, 30 minutes, and 1, 2, 4, 8, 12, 24, 48, 72, and 96 hours, and 14 days after the beginning of EXPAREL administration
Time Frame: Baseline, 0.25, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, and 96 hours, and 14 days post-dose
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | Bupivacaine FNB + EXPAREL Infiltration | Bupivacaine FNB + EXPAREL Infiltration Admixed With Bupivacaine
Number analyzed (Participants) | 6 | 1
hours*ng/mL | 25134 (11506) | 38489 (NA)

5. Primary Outcome: The Apparent Terminal Elimination Rate Constant (λz)
Description: Blood samples for bupivacaine PK analysis were to be obtained from subjects at baseline (prior to bupivacaine HCl administration for nerve block), 15 minutes, 30 minutes, and 1, 2, 4, 8, 12, 24, 48, 72, and 96 hours, and 14 days after the beginning of EXPAREL administration
Time Frame: Baseline, 0.25, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, and 96 hours, and 14 days post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/hours
Arm/Group | Bupivacaine FNB + EXPAREL Infiltration | Bupivacaine FNB + EXPAREL Infiltration Admixed With Bupivacaine
Number analyzed (Participants) | 6 | 1
1/hours | 0.0290 (0.0089) | .0315 (NA)

6. Primary Outcome: The Apparent Terminal Elimination Half-life (t1/2el)
Description: as for outcome 5
Time Frame: Baseline, 0.25, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, and 96 hours, and 14 days post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Bupivacaine FNB + EXPAREL Infiltration | Bupivacaine FNB + EXPAREL Infiltration Admixed With Bupivacaine
Number analyzed (Participants) | 6 | 1
hours | 25.9 (8.02) | 22 (NA)

ADVERSE EVENTS:
Time Frame: Adverse events were to be monitored from the time the informed consent form was signed through Day 14 post-dose.
Groups:
- Bupivacaine FNB + EXPAREL Infiltration Admixed With Bupivacaine: Femoral nerve block (FNB) with bupivacaine HCl 0.5% with epinephrine 1:200,000 within 2 hours of the surgical procedure. Infiltration of EXPAREL 266 mg admixed with bupivacaine HCl 0.5% with epinephrine 1:200,000 just prior to wound closure.
  Bupivacaine FNB: A single administration of bupivacaine HCl 0.5% with epinephrine 1:200,000 in 20 mL volume will be administered within 2 hours prior to the surgical procedure as an ultrasound-guided FNB.
  EXPAREL Infiltration: A single dose of EXPAREL 266 mg expanded to 60 mL with preservative-free sterile normal saline admixed with bupivacaine HCl 0.5% with epinephrine 1:200,000 infiltrated into the surgical site just prior to wound closure.
Arm/Group | Bupivacaine FNB + EXPAREL Infiltration | Bupivacaine FNB + EXPAREL Infiltration Admixed With Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/7
Other Adverse Events (participants affected / at risk) | 1/16 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine FNB + EXPAREL Infiltration (N=16) | Bupivacaine FNB + EXPAREL Infiltration Admixed With Bupivacaine (N=7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No